CLINICAL TRIAL: NCT06144034
Title: Effect of Air Polishing for Biofilm Removal on Clinical, Biological, and Patient-Reported Experience Among Epileptic and Non-Epileptic Children: A Split-Mouth Randomised Clinical Trial
Brief Title: Air Polishing Effect on Biological, Clinical and Patient-reported Experience Among Epileptic and Non-epileptic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 635-2022
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy; Gingivitis
Keywords: Air polishing; Airflow; Erythritol; Oral health of special healthcare needs children
MeSH Terms: conditions — Epilepsy; Gingivitis | interventions — Pulmonary Ventilation

STUDY DESIGN:
Intervention Model Description: Split-Mouth Design Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor was blinded to treatment intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epilepsy patients (Experimental): 1 and 3 quadrants got the same treatment and 2 and 4 got the same treatment. Air polishing with erythritol powder was used to remove biofilm and EMS ultrasonic scaler to remove calculus if present. also rubber cup and prophylaxis paste spearmint (Kemdent Works, Purton. Swindon, Wiltshire. SN5 4HT, UK). and EMS ultrasonic scaler to remove calculus if present.
  Interventions: Device: Air polishing with erythritol powder; Device: Conventional treatment
- Non-epileptic pateints (Experimental): 1 and 3 quadrants got the same treatment and 2 and 4 got the same treatment. Air polishing with erythritol powder was used to remove biofilm and EMS ultrasonic scaler to remove calculus if present. also rubber cup and prophylaxis paste spearmint (Kemdent Works, Purton. Swindon, Wiltshire. SN5 4HT, UK). and EMS ultrasonic scaler to remove calculus if present.
  Interventions: Device: Air polishing with erythritol powder; Device: Conventional treatment

INTERVENTIONS:
Device: Air polishing with erythritol powder — Air polishing with erythritol powder utilized for biofilm disclosing and, followed by an ultrasonic scaler to remove calculus if present.
  Other Names: Airflow
Device: Conventional treatment — Rubber cup polishing with prophy paste after biofilm disclosing, followed by ultrasonic scaling of calculus if present.
  Other Names: Rubber cup polishing

SUMMARY:
In epileptic and non Epileptic children, the full dentition of each patient was split into four quadrants, starting from the upper right quadrant (1) and moving clockwise until the lower right quadrant (4). Bundled into two groups: quadrant (1+3) vs. (2+4). After randomization, each of these pairs of quadrants had the same treatment modality; test quadrants received treatment with airflow to remove soft biofilm, and ultrasonic scaler for areas with calculus deposits, and control quadrants were treated with conventional rubber cup polishing to remove soft biofilm and ultrasonic scaler for calculus deposits.

DETAILED DESCRIPTION:
The treatment of each quadrant was administered sequentially, beginning with the upper right quadrant. Treatment duration was measured in seconds from the start of treatment in each quadrant until the removal of all disclosed biofilm and calculus. This process was repeated for each quadrant individually. And intra-oral photographs were taken before, immediately after treatment, and at follow-up time.

Conventional treatment was conducted after biofilm disclosure by a rubber cup and prophylaxis paste spearmint (Kemdent Works, Purton. Swindon, Wiltshire. SN5 4HT, UK). The power setting was between 70% and 100%. The rubber cup was used until all biofilm was removed, then, if present, calculus was removed by Electro Medical Systems (EMS) ultrasonic scaler with a power setting between 3-6 on the Airflow control panel.

For Airflow, treatment was conducted after biofilm disclosure. The powder chamber of the air polishing device was filled with low-abrasive erythritol powder, according to the manufacturer's instructions. The tip of the handpiece was positioned at an angle of 70° to the surface of the tooth to be polished at 3 mm from the tooth surface. Once activated, a non-stop movement from mesial to distal and distal to mesial in a smiley face shape starting from the gingival sulcus and moving upwards coronally to the incisal to cover the entire clinical crown was performed, with a power setting ranging from 3-6 on the control panel of the airflow device. EMS ultrasonic scaler was used to remove calculus if present with a power ranging from 3-6.

ELIGIBILITY:
Inclusion Criteria:

* children aged 5 to 15 years with epilepsy
* on anti-epileptic drugs (AED) for at least 3 months
* periodontal pockets depths not exceeding 3mm
* full-mouth plaque scores over 50%, and having 5 teeth per quadrant.
* The non-epileptic group included healthy non-epileptic children meeting similar criteria for age, periodontal health, and plaque scores

Exclusion Criteria:

* coexisting neurological illnesses other than epilepsy, medical conditions impacting oral health, periodontitis, asthma, swallowing difficulties, intellectual disabilities, and non-ambulatory status

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Gingival inflammation | Before treatment began, and two weeks after treatment.
  using Loe and Silness gingival index. Before biofilm disclosing, evaluated by assigning scores from 0-3 for gingival inflammation at four sites (mesial, distal, buccal, and lingual/palatal) per tooth, 0- normal gingiva and 3 - severely inflamed
Mean Marginal Plaque | Before treatment began, immediately after, and two weeks after treatment.
  O'Leary Plaque Index on 6 sites per tooth, 0= absence of plaque or 1= presence of plaque
patient satisfaction | immediately after treatments of each quadrant.
  Likert Faces 5-points satisfaction scale, 0-4, 0 = Very dissatisfied. 4= Very satisficed
Treatment duration | from the time procedure begins until removing all dental biofilm and calculus
  for each quadrant, time was measured from beginning of treatment till biofilm and calculus are fully removed per seconds
Pain measure | immediately after treatments of each quadrant.
  Faces pain scale-Revised 0-10, 0 no pain, 10 maximum pain
patient satisfaction | immediately after treatments of each quadrant.
  two questions, Which treatment method was less painful, Which treatment would you do again?

SECONDARY OUTCOMES:
Biomarkers | Before treatment began, and two weeks after treatment.
  Gingival crevicular fluid samples IL-1B and MMP-8 two samples per patient, one for each treatment method
Residual plaque area | Before treatment began, immediately after, and two weeks after treatment.
  Rustogi modified Navy plaque index

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - Jordan Univerity of Science and technology, Irbid
  - Jordan University of Science and Technology, Irbid